CLINICAL TRIAL: NCT04597073
Title: Measurement of Oncostatin M, Leukemia Inhibitory Factor and Interleukin-11 Levels in Serum, Saliva, and Gingival Crevicular Fluid of Patients With Periodontal Disease
Brief Title: Measurement of Oncostatin M, Leukemia Inhibitory Factor and Interleukin-11 Levels of Patients With Periodontal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Tugba Aydin, Assistant Professor, Ataturk University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: OncosM,LIF,IL-11
Record Dates: First submitted 2020-10-06; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Chronic Periodontitis, Generalized; Gingivitis
Keywords: Chronic Periodontitis; Gingival Crevicular Fluid; Leukemia Inhibitory Factor; Oncostatin M; Interleukin-11; Periodontal Therapy; Gingivitis
MeSH Terms: conditions — Chronic Periodontitis; Gingivitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy (No Intervention): included individuals with probing depth (PD) ≤3mm, no sites with attachment loss, and no radiographic evidence of alveolar bone resorption. They exhibited no sign of inflammation (GI=0).
- Gingivitis (Experimental): had varying degrees of gingival inflammation (GI≥1), PD≤3mm with no clinical attachment loss or with no alveolar bone destruction.
  Interventions: Procedure: Initial Periodontal Therapy
- Chronic Periodontitis (Experimental): was defined as those who were with PD ≥ 4mm, clinical attachment loss (CAL) ≥ 2mm, and who had bone loss affecting >30% of the existing teeth on clinical and radiographic examination.
  Interventions: Procedure: Initial Periodontal Therapy

INTERVENTIONS:
Procedure: Initial Periodontal Therapy — Oral hygiene education, including the use of toothbrushes and dental floss and/or interproximal brushes, was given to them. After one week Chronic Periodontitis group received nonsurgical periodontal therapy consisting of scaling and root planing (quadrant by quadrant) using manual scalers and curettes under local anesthesia. No antibiotics or any medications were prescribed during the treatment. Periodontal treatment was performed by the same investigator
  Arms: Chronic Periodontitis; Gingivitis

SUMMARY:
This study aims to determine Oncostatin M (OSM), Leukemia inhibitory factor (LIF), and Interleukin-11 (IL-11) levels in gingival crevicular fluid (GCF), saliva, and serum in periodontally healthy individuals and those with gingivitis and chronic periodontitis before and after periodontal treatment and to evaluate the relationship between these cytokine levels and clinical periodontal parameters.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy
* non-smokers

Exclusion Criteria:

* smokers
* pregnancy or lactation
* individuals with any systemic disease
* individuals who have had periodontal treatment in the last six months

Ages: 20 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level baseline | baseline (before treatment)
  As described by Silness&Löe 1964; The measurement of the state of oral hygiene by Silness-Löe plaque index is based on recording both soft debris and mineralized deposits on the following teeth. Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3. Scores 0: No plaque. scores 1: A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  Scores 2: Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye.
  Scores 3: Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  Score 0 considered good oral hygiene, score 3 bad oral hygiene habits. plaque index for a tooth=scores from 4 areas/4 plaque index individual= scores from 28 tooth/28
Plaque index baseline | baseline (before treatment)
  As described by Silness&Löe 1964; The measurement of the state of oral hygiene by Silness-Löe plaque index is based on recording both soft debris and mineralized deposits on the following teeth. Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3.
  Scores 0: No plaque. scores 1: A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  Scores 2: Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye.
  Scores 3: Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  Score 0 considered good oral hygiene, score 3 bad oral hygiene habits. plaque index for a tooth=scores from 4 areas. plaque index individual= scores from 28 tooth
Gingival index baseline | baseline (before treatment)
  As described by Löe&Silness 1963; The bleeding is assessed by probing gently along the wall of soft tissue of the gingival sulcus. Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3.
  Score 0 - Normal, healthy gingival with sharp, non-inflamed margins. score 1 - Marginal gingivitis with minimal inflammation and edema at the free gingival. No bleeding on probing.
  Score 2 - Moderate gingivitis with a wider band of inflammation and bleeding upon probing.
  Score 3 - Advanced gingivitis with inflammation clinically reaching the mucogingival junction usually with ulceration.
  Score 0 considered healthy gingiva, score 3 assessed advanced gingival disease. gingival index for a tooth=scores from 4 areas/4 gingival index individual= scores from 28 tooth/28
Probing of depth baseline | baseline (before treatment)
  Measurement to the nearest millimeter from the gingival margin to the base of the clinical pocket by Williams periodontal probe
Biochemical outcomes baseline | baseline (before treatment)
  In this study, biochemical parameters including OSM,LIF, IL-11 were measured (pg/ml) by ELISA (Enzyme-Linked Immuno Sorbent Assay) measured (pg/ml) by ELISA (Enzyme-Linked Immuno Sorbent Assay) methods on Gingival Crevicular Fluid, saliva and serum at baseline

SECONDARY OUTCOMES:
Clinical attachment level after 8 weeks | 8 weeks after treatment
  Calculation as distance in millimeters from cement-enamel junction to the bottom of the pocket by Williams periodontal probe
Plaque index after 8 weeks | 8 weeks after treatment
  As described by Silness&Löe 1964; The measurement of the state of oral hygiene by Silness-Löe plaque index is based on recording both soft debris and mineralized deposits on the following teeth. Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3.
  Scores 0: No plaque scores 1: A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  Scores 2: Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye. Scores 3: Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  Score 0 considered good oral hygiene, score 3 bad oral hygiene habits. plaque index for a tooth=scores from 4 areas/4 plaque index individual= scores from 28 tooth/28
Gingival index after 8 weeks | 8 weeks after treatment
  As described by Löe&Silness 1963; The bleeding is assessed by probing gently along the wall of soft tissue of the gingival sulcus. Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3.
  Score 0 - Normal, healthy gingival with sharp, non-inflamed margins. score 1 - Marginal gingivitis with minimal inflammation and edema at the free gingival. No bleeding on probing. Score 2 - Moderate gingivitis with a wider band of inflammation and bleeding upon probing.
  Score 3 - Advanced gingivitis with inflammation clinically reaching the mucogingival junction usually with ulceration.
  Score 0 considered healthy gingiva, score 3 assessed advanced gingival disease. gingival index for a tooth=scores from 4 areas/4 gingival index individual= scores from 28 tooth/28
Probing of dept after 8 weeks | 8 weeks after treatment
  Measurement to the nearest millimeter from the gingival margin to the base of the clinical pocket by Williams periodontal probe
Biochemical outcomes after 8 weeks | 8 weeks after treatment
  In this study, biochemical parameters including OSM,LIF, IL-11 were measured (pg/ml) by ELISA (Enzyme-Linked Immuno Sorbent Assay) measured (pg/ml) by ELISA (Enzyme-Linked Immuno Sorbent Assay) methods on Gingival Crevicular Fluid, saliva and serum at 8 weeks